CLINICAL TRIAL: NCT00262418
Title: A Randomised, Double Blind, Double Dummy Study to Compare the Efficacy and Safety of a Single Administration of Ivermectin to a Single Administration of Permethrin for the Treatment of Scabies
Brief Title: Comparison of the Efficacy and Safety of Ivermectin to Permethrin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2004/212
Record Dates: First submitted 2005-12-04; First posted 2005-12-06 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies | interventions — Permethrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of ivermectin or permethrin

SUMMARY:
Comparison of the efficacy and safety of a single administration of ivermectin to a single administration of permethrin for the treatment of scabies

DETAILED DESCRIPTION:
Administration of ivermectin or permethrin on day0 Clinical examination and pictures on day0, day14 and day28 Blood sample on day0 VAS for pruritus, DLQI and SF-36 on day0, day14 and day28

ELIGIBILITY:
Inclusion Criteria:

At least one of the following inclusion criteria:

* Scabies tunnels
* Positive microscopic examination (acarids, faeces or ova)

At least two of the three following inclusion criteria:

* Non-specific injuries with a typical distribution pattern
* Serious itching which increases during the night
* Family or contacts with similar complaints

Exclusion Criteria:

* Treatment for scabies < 4 weeks ago
* Treatment with corticoids < 1 week ago
* Pregnancy
* Breast-feeding
* HIV
* Serious immunodepressive patients
* Sensitivity or allergy to one of the components of the study medication
* Damage of the central nerve system

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-07; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Clinical healing of the skin injuries | on day28

SECONDARY OUTCOMES:
Decrease of itching | on day28
Amelioration of the life quality | on day28
Number and gravity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Naeyaert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be